CLINICAL TRIAL: NCT00741130
Title: Corrected Measurement of the Retinal Nerve Fiber Layer Thickness by Optic Disc Configuration With the Cirrus HD OCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Gong Je Seong, Yonsei University College of Medicine
Other Study IDs: 3-2008-0076
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 2008-08

CONDITIONS: Glaucoma; Myopia
Keywords: retinal nerve fiber layer; optic nerve head; Cirrus OCT
MeSH Terms: conditions — Glaucoma; Myopia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- C: normal volunteers
- G: glaucoma patients

SUMMARY:
Because the measurement of the retinal nerve fiber layer thickness is very sensitive to the position of measurement, it may be incorrect in patients with the tilted disc. In the present study, the corrected RNFL thickness by the optic nerve head configuration using the Cirrus HD OCT will be evaluated. If the corrected RNFL thickness is more sensitive to detect the localized RNFL defect, the present software should be upgrade to reflect the optic nerve head configuration.

DETAILED DESCRIPTION:
Finding the localized retinal nerve fiber layer (RNFL) defect and measuring the RNFL thickness are two main issues for early glaucoma detection. A recently developed imaging device, the Cirrus HD OCT, offers more detailed informations about retina architecture including optic nerve head. To calculate the RNFL thickness, the software of the Cirrus HD OCT supposes an ideal optic nerve head. However, in the cases with not ideal optic disc configuration, the measurement of the RNFL thickness is not correct. Because the measurement of the RNFL thickness is extremely sensitive to the position of measurement, patients with the tilted disc are in danger of misdiagnosis. In the present study, we want to correct the RNFL thickness measurement according to the optic nerve head configuration using the Cirrus HD OCT. If the corrected RNFL thickness is more sensitive to detect the localized RNFL defect, the present software should be upgrade to reflect the optic nerve head configuration.

ELIGIBILITY:
Inclusion Criteria:

* normal controls or glaucoma patients
* signal intensity of the OCT image > 8
* cooperative subjects

Exclusion Criteria:

* spherical equivalent refractive errors > +4 diopters or < -4 diopters
* significant media opacity
* previous intraocular surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers of our opthalmologic clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-10 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
the Cirrus HD OCT | when the OCT images are taking

SECONDARY OUTCOMES:
automated visual field | when the OCT images are taking
red-free fundus photo | when the OCT images are taking
refractive errors | when the OCT images are taking

CONTACTS AND LOCATIONS:
Overall Officials: Gong Je Seong, MD, PhD, Study Chair — Yonsei University
Locations (1):
- Gong Je Seong, Seoul, South Korea